CLINICAL TRIAL: NCT04388696
Title: A Gender Transformative Program to Prevent Sexual Violence and Relationship Abuse Among Adolescent Women: A Feasibility Trial of Sisterhood 2.0
Brief Title: A Feasibility Trial of Sisterhood 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Department Human Services, Pennsylvania (Unknown); Fisa Foundation (Unknown); The Grable Foundation (Unknown)
Responsible Party: Principal Investigator, Elizabeth Miller, Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO17010174
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Adolescent Behavior; Violence in Adolescence; Group, Peer; Violence, Non-accidental; Violence, Sexual; Violence, Physical; Violence, Domestic; Emotional Abuse; Coping Skills; Communication, Personal
MeSH Terms: conditions — Adolescent Behavior; Coitus; Communication

STUDY DESIGN:
Intervention Model Description: The 18-24 hour content (divided into 8, 3 hour sessions) are spread over a 3 week to 2 month period. Sessions explored gender, consider harmful messages around femininity and socially acceptable images of women, healthy sexuality, healthy relationships and connections, understanding and identifying sexual abuse and assault, and self care.
  Control Program: The control intervention used widely-used curricula focused on job skills development and life skills. Trained prevention educators provided the programs for both intervention and control arms and were trained to implement either the Sisterhood 2.0 program or the job skills curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sisterhood 2.0 (Experimental): Sisterhood 2.0 used a group format with activities that explore respect, nonviolence, healthy relationships, and sexuality, through 8 sessions (3 hours/session) over an 8 week period.
  Sessions focus on gender, consider harmful messages around femininity and their image, healthy sexuality, healthy relationships and connections, understanding sexual abuse and assault, and self care.
  Interventions: Behavioral: Sisterhood 2.0
- Job Skills Training (Active Comparator): The curriculum used for this program is an intensive 18-24 hour job readiness training curriculum distributed across 3 weeks, or up to 2 months.
  Interventions: Behavioral: Sisterhood 2.0

INTERVENTIONS:
Behavioral: Sisterhood 2.0 — The Sisterhood 2.0 curriculum was adapted from Program M, created in 2006 by Promundo to address health and empowerment of young women aged 15-24. The curriculum engages young women in questioning rigid and non-equitable stereotypes about masculinity and femininity and how they affect both women's and men's health and well-being.

SUMMARY:
This pilot quasi-experimental community based trial examines the feasibility of a sexual violence and adolescent relationship abuse prevention program for girls aged 14-19. Feasibility is assessed through participant attendance, retention and program satisfaction measures and interviews are conducted at baseline, end of program and 3 month follow up (endline) about participant experiences.

DETAILED DESCRIPTION:
The goal of the project is to adapt and pilot a "gender transformative," sexual violence and adolescent relationship abuse prevention program, Sisterhood 2.0, among African American high school-age females in a community-based setting. The Sisterhood 2.0 curriculum was adapted from Program M, created in 2006 by Promundo to address health and empowerment of young women aged 15-24. The curriculum engages young women in questioning rigid and non-equitable stereotypes about masculinity and femininity and how these rigid stereotypes affect their health and well-being. This study will pilot test, using a quasi-experimental design, the participant satisfaction with the program through measures of attendance and retention, and be compared to a job skills development curriculum. This study is significant because there are too few evidence-based sexual violence and adolescent relationship abuse prevention program in the U.S., none that are specifically tailored for African American adolescent females, and there are no evidence- based programs implemented in community settings that target both sexual violence and adolescent relationship abuse and adolescent sexual health.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ages 13-19 (inclusive)
* Participants must speak English
* Participants must self identify as female

Exclusion Criteria:

* Not ages 13-19 (inclusive)
* Does not speak English
* Does not identify as female

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self identifying females aged 13-19.
Enrollment: 246 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Participant Attendance | through study completion, an average of 1 per week
  Attendance recorded at beginning and end of each session with a weekly satisfaction survey. Calculated as a proportion of total number of sessions.
Participant Retention | post-intervention at Week 8
  At the end of the program, participants were asked why they returned or did not return to the program each week and their reasons for missing any sessions.
Participant Satisfaction | through study completion, an average of 1 per week
  Participants were asked about how satisfied they were with the topic discussed and format of the program each week.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The research team will not make individual participant data (IPD) available to other researchers. This plan to Share IPD is consistent with the IPD Sharing Plan Description for our collaborating agency.